## **Statistical Analysis Plan**

## **Study Title:**

Developing a Low-Intensity, Primary Care Intervention for Anxiety Disorders

**Date:** 7/17/2017

**NCT#:** NCT02579915

We established a priori benchmarks for feasibility, acceptability, and preliminary efficacy for this treatment development project. For efficacy, the benchmark was: at least 50% of participants experience a 20% reduction in HARS. In the RCT, 63% (5/8) of participants randomly assigned to the intervention who completed the post-treatment assessment met our HARS benchmark compared to 38% (6/16) in the symptom monitoring control condition.